CLINICAL TRIAL: NCT01889147
Title: A Single Dose Study to Assess the Peak Plasma Concentration of a Microdose of Recombinant Human Placental Alkaline Phosphatase (hRESCAP, Part 1) Followed by a Single Ascending Dose, FIH Study to Assess Safety and Tolerability of hRESCAP (Part 2).
Brief Title: Microdose and First-In-Human (FIH) Study of Recombinant Human Placental Alkaline Phosphatase (hRESCAP)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Alloksys Life Sciences B.V. (Industry)
Responsible Party: Principal Investigator, W.J. Pasman, Project Manager Clinical Studies Food and Pharma, TNO
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CHDR1220
Record Dates: First submitted 2013-06-18; First posted 2013-06-28 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Peak plasma concentration; safety and efficacy; therapeutic agent; LPS-mediated diseases; Pharmacokinetics of administered hRESCAP; Determine half-time

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 14C-hRESCAP (Active Comparator): Peak plasma concentration response of a dose hRESCAP will be examined and compared with the saline condition
  Interventions: Biological: hRESCAP
- saline (Placebo Comparator): Peak plasma concentration response of different dosages of hRESCAP will be examined and controlled with the saline condition
  Interventions: Biological: Placebo
- Microdose (Active Comparator): Peak plasma concentration of a very low dose of hRESCAP as a first test in humans (first starting dose, before the other arms).
  Interventions: Biological: hRESCAP

INTERVENTIONS:
Biological: hRESCAP — one acute bolus administration of different dosages of hRESCAP (microdose, part 1; and FIH: low dose, 414 µg; medium dose, 2480 µg; high dose, 5300 µg; part 2)
  Other Names: recombinant human placental alkaline phosphatase
  Arms: 14C-hRESCAP; Microdose
Biological: Placebo
  Arms: saline

SUMMARY:
In the present study human recombinant placental alkaline phosphatase (hRESCAP) will be investigated. Alkaline Phosphatase is naturally present in the body and reported to use lipopolysaccharde (LPS, bacterial endotoxins) and extracellular nucleotides leaking from damaged and ischemic cells as physiological substrates. The LPS-substrate prevalence makes alkaline phosphatase an interesting novel therapeutic agent in the treatment of LPS-mediated diseases. A bovine homologue of this protein (bovine intestinal alkaline phosphatase, BIAP) has previously been investigated for treatment of acute inflammatory responses such as sepsis, and was shown to be safe in humans. hRESCAP, which will be investigated in the current study, is expected to have a longer half-life in humans than the previously investigated BIAP, due to the fact that it is more sialylated. The possibility to increase the t1/2 to days instead of minutes enables treatment of chronic diseases.

DETAILED DESCRIPTION:
In the current study the peak plasma concentration (pharmacokinetics/elimination) of [14C]-labelled hRESCAP in healthy volunteers will be investigated at increasing single doses (up to anticipated therapeutic dose), with a microdose (≤30 nmol) as a safe starting dose.

* Part 1: To assess the peak plasma concentration of a single microdose (≤30 nmol) of a recombinant human protein (hRESCAP), administered intravenously, as a suitable technique to predict the pharmacokinetics in humans at pharmacologically relevant doses;
* Part 2: To determine the safety and tolerability of single dose of hRESCAP up to 5300 µg in healthy male volunteers administered intravenously;
* To determine the peak plasma concentration of hRESCAP in healthy male volunteers within a pharmacologically relevant dose-range and compare this with BIAP pharmacokinetics with emphasis on half-life (t1/2).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, 18 - 45 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, haematology, blood chemistry, and urinalysis;
2. Body mass index (BMI) between 18 and 30 kg/m2, inclusive;
3. Ability to communicate well with the investigator in the Dutch language;
4. Able to participate and willing to give written informed consent and to comply with the study restrictions;
5. Venous access sufficient to allow blood sampling as per protocol.

Exclusion Criteria:

1. Any clinically significant abnormality as determined by medical history taking and physical examinations obtained during the screening visit that in the opinion of the investigator would interfere with the study objectives or compromise subject safety;
2. History of a surgical event that may significantly affect the study outcome;
3. History of allergy or other inflammatory indications;
4. History of asthma or other inflammatory disease;
5. Use of prescription medications, over the counter medications, vitamin, herbal and dietary supplements within 21 days prior to study drug administrations, or less than 5 half-lives, whichever is longer, and during the course of the study.
6. Alkaline Phosphatase levels in plasma of < 30 IU/L or > 115 IU/L;
7. Clinically relevant abnormal laboratory results, ECG, vital signs, or physical findings at screening that in the opinion of the investigator would interfere with the study objectives or compromise subject safety;
8. Participation in an investigational drug, food (ingredients) or device study within 3 months prior to screening or more than 4 times in the past year;
9. Any psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol;
10. History of alcohol or illicit drug abuse (alcohol abuse defined as alcohol consumption > 28 units/week);
11. Reported unexplained weight loss or weight gain of > 2 kg in the month prior to screening;
12. Positive test results for Hepatitis B, Hepatitis C or HIV;
13. Donation of blood within 3 months prior to screening or donation of plasma within 14 days prior to screening;
14. Not having a general practitioner;
15. Not willing to accept information transfer which concerns participation in the study, or information regarding health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner;
16. Not willing to give permission to have the general practitioner to be notified upon participation in this study;
17. Prior participation in part 1 is not allowed for subjects participating in part 2.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the peak plasma concentration of hRESCAP after microdose administration of hRESCAP | 35 days
  After administration of hRESCAP intravenously, blood will be withdrawn of the subjects frequently for in total 35 days (five times the anticipated half-life period of one week).

SECONDARY OUTCOMES:
In the ascending dose study increased dosages of of hRESCAP will be supplied till finally the therapeutic dose. | Two weeks (based upon time phrame of micodose section of the study)
  In three subjects a low, medium and high dose of hRESCAP will be administered and a control saline administration in one subject. The peak plasma concentration of hRESCAP response of different dosages will be useful for treatment evaluation. The administration of the different dosages supplied is one week apart for safety reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Koos Burggraaf, MD, PhD, Principal Investigator — CHDR
Locations (1):
- Centre for Human Drug Research, Leiden, South Holland, Netherlands